CLINICAL TRIAL: NCT04023383
Title: The Effect of New Cross Linked Hyaluronan Gel on Quality of Life of Patients After Deep Infiltrating Endometriosis Surgery: A Randomized Controlled Pilot Study
Brief Title: New Cross Linked Hyaluronan Gel After Deep Infiltrating Endometriosis Surgery
Acronym: HYALOENDOQoL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HYALOENDOQoL
Record Dates: First submitted 2019-07-13; First posted 2019-07-17 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Endometriosis; Adhesion; Quality of Life; Surgery
MeSH Terms: conditions — Endometriosis; Tissue Adhesions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): The patients in the control group had 40 cc sterile saline solution compatible with the body temperature.
  Interventions: Drug: 40 cc sterile saline solution
- HyaRegen NCH gel group (Experimental): In the intervention group had 40 mL of HyaRegen NCH gel instilled into the peritoneal cavity through a large-bore cannula following standard laparoscopic procedures.
  Interventions: Drug: 40 cc HyaRegen NCH gel

INTERVENTIONS:
Drug: 40 cc HyaRegen NCH gel — After an extensive bleeding control the patients in the intervention group had 40 mL of HyaRegen NCH gel instilled into the peritoneal cavity.
  Other Names: bleeding control
  Arms: HyaRegen NCH gel group
Drug: 40 cc sterile saline solution — After an extensive bleeding control the patients in the control group had 40 cc sterile saline solution compatible with the body temperature.
  Other Names: bleeding control
  Arms: Control

SUMMARY:
Hyaluronan, a glycosaminoglycan found in connective tissues and extracellular matrix, has been postulated to reduce postoperative adhesions, because of its unconditioned biological functions at tissue repair but unfortunately it has a fluid nature that causes rapid degradation, and it cannot effect long enough to work as an adhesion barrier.(10,11) For this reason a New cross-linked hyaluronan (NCH) gel, that has higher viscosity compared to natural hyaluronan has been developed by BioRegen Biomedical (Changzhou, Jiangsu, China). It has the ability for gradually absorption within 1 to 2 weeks in vivo, which are the acquired repair period and the critical time for adhesion formation. Although it seems evident that endometriosis has a serious impact on the daily Quality of Life of women; comparable data for the effect of adhesion barriers to patients who have had laparoscopic (Deep infiltrating endometriosis) DIE surgery is missing.

Therefore a pilot randomised controlled study was conducted to evaluate the effect of NCH gel on short term quality of life in patients who had undergone laparoscopic surgery due to DIE.

DETAILED DESCRIPTION:
A prospective 1:1 randomised placebo-controlled study was conducted in our department during the study period January 2017-January 2019. All patients were included after obtaining written, signed informed consent before participating. All of the procedures were performed by the same surgery team who are experienced in minimally invasive (Deep infiltrating endometriosis) DIE surgery. The study protocol was approved by the local Ethics Committee of hospital (Approval number: 2017/04/35) 60 patients who were underwent for laparoscopic surgery for the treatment of deep infiltrating endometriosis without bowel involvement were recruited.

The inclusion criteria for this study were as follows, aged 18 to 45 years, and undergoing laparoscopic surgery for suspicious of DIE and persistent pain irrespective to any medical treatment. Patients were booked for follow-up visits at the 3rd and 6th month postoperative months and wanted to fill the questionnaires.

The exclusion criteria for the study were as; acute or severe infection, autoimmune disease, known/suspected intolerance or hypersensitivity to Hyaluronan or its derivatives, concurrent use of a systemic anti-inflammatory or hormonal drug at least 3 months prior to the surgery, clinical evidence of cancer; use of anticoagulant, fibrin glue, other thromboembolic agents, or any other anti-adhesion agent during the procedure ,patients with surgically diagnosed bowel involvement or need bowel resection, and who want to receive any postoperative hormonal treatment.

Participants were allowed to voluntarily withdraw from the trial for any reason at any time, and could be terminated by investigators owing to safety concerns, violations of inclusion/exclusion criteria, or pregnancy.

Surgical procedure The patients were laid low lithotomy position under general anesthesia. Patients were assigned at random to either the NCH gel or control group in a 1:1 ratio through a computer based program. A standardised technic with 4 abdominal incision laparoscopic approach with 10 mm umbilical trocar for the optic camera and three 5 mm axillary ports for the surgical instruments were used. All of the surgeries initiated from exploring the pelvic cavity, identification of the ureters and dissection transection of the pelvic adhesion by 5 mm bipolar cautery used at 25 kw for coagulation mode and scissors. The incision was begun on the left pelvic sidewall just cephalad to the last deposit. The incision was then extended towards the uterus, lateral and parallel to the left uterosacral ligament. The uterosacral ligament was pushed medially and down and the healthy tissues including the ureter were pushed upwards and laterally away from the dissection. It then transected the right utero-sacral ligament and was continued along the right pelvic sidewall just lateral and above the right uterosacral ligament until it extends beyond all obvious deposits. All of the endometriotic foci was grasped and pulled then undercut and freed so that the whole lesion and a surrounding margin of healthy tissue was removed. After an extensive bleeding control the Patients in the intervention group had 40 mL of HyaRegen NCH gel instilled into the peritoneal cavity through a large-bore cannula following standard laparoscopic procedures. The patients in the control group had 40 cc sterile saline solution compatible with the body temperature. Operators could not be blinded to treatment allocation, but the questionnaire assessors and the patients were blinded to treatment allocation.

Pre and Postoperative assessment of pain and quality of life A dedicated research assisted in this study was asked the validated (visual analogue scale) VAS (dysmenorrhea, dyschezia, dyspareunia, dysuria, and pelvic pain), (endometriosis health profile-5) EHP-5 and (short form 12) SF-12 questionnaires before the day of the surgery. (12-14) A validated form of VAS score was used and scored from 0: No pain to 10: the worst pain all in their lives in a likert fashion. The VAS and (quality of life ) QoL questions were asked then in the 3rd and 6th month of during their follow up visits. A validated form of SF-12 that includes physical functioning, role limitation due to physical health problems, bodily pain, general health, vitality (energy/fatigue) social functioning, role limitations due to emotional problems and mental health (psychological distress or wellbeing) were asked. The questions are scored and analysed using a statistical algorithm to give two scores: the physical component summary and the mental component summary.

A validated form of EHP-5 questionnaire was used to determine endometriosis related QoL of the patients. EHP-5 consists of two parts: the first has a central questionnaire that evaluate five dimensions - pain, control and powerlessness, emotional well-being, social support, and self-image; and the second part measuring the areas of sexual intercourse, work, relationship with children, feelings about medical professional, treatment and infertility.

Statistical analysis Data analysis was performed by using SPSS (IBM SPSS Statistics for Windows, Version 20.0. Armonk, NY: IBM Corp.). A one-sample Kolmogorov-Smirnov test was performed to analyse the distribution of clinical variables. The frequency and percentage of the categorical variables and the mean, standard deviation, median and range values of the continuous and ordinal variables were presented. The study groups were compared using Student t test for parametric variables and Mann Whitney U test for the non-parametric variables. A post-hoc sample size calculation was performed via a two-sided Z test (α=0.05, β=0.20) for each study groups in order to obtain VAS scores as the primary outcome A p-value of < 0.05 was considered statistically significant for all calculations

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 45 years
* undergoing laparoscopic surgery for suspicious of DIE
* persistent pain irrespective to any medical treatment

Exclusion Criteria:

* acute or severe infection
* autoimmune disease
* known/suspected intolerance or hypersensitivity to hyaluronan or its derivatives
* concurrent use of a systemic anti-inflammatory or hormonal drug at least 3 months prior to the surgery
* clinical evidence of cancer
* use of anticoagulant, fibrin glue, other thromboembolic agents
* use of any other anti-adhesion agent during the procedure
* patients with surgically diagnosed bowel involvement or need bowel resection
* patients who want to receive any postoperative hormonal treatment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
The preoperative and postoperative 3rd and 6th month change of Visual Analogue Scale symptom score | The preoperative and postoperative 6th month change in Visual Analogue Scale symptom score
  A validated form of VAS score was used and scored from 0: No pain to 10: the worst pain all in their lives in a likert fashion.

SECONDARY OUTCOMES:
Short Form-12 Quality of Life | The preoperative and postoperative 3rd and 6th month change of Short Form-12 Quality of Life questions were recorded considering follow up visits.
  A validated form of Short Form-12 Quality of Life that includes physical functioning, role limitation due to physical health problems, bodily pain, general health, vitality (energy/fatigue) social functioning, role limitations due to emotional problems and mental health (psychological distress or wellbeing) were asked. The scores may be reported as Z-scores (difference compared to the population average, measured in standard deviations). We used an online programme (https://www.orthotoolkit.com/sf-12) to calculate Short Form-12 Quality of Life total and sub-scale results. The maximum PCS-12 (Physical Score) is 55.57 and the maximum MCS-12 (Mental Score) is 60.75. The minimum PCS-12 (Physical Score) is 22.99 and the minimum MCS-12 (Mental Score) is 19.06.
Endometriosis Health Profile (EHP-5) | The preoperative and postoperative 3rd and 6th month change of A validated form of
  A validated form of Endometriosis Health Profile (EHP-5)

CONTACTS AND LOCATIONS:
Overall Officials: Murat Ekin, MD, Principal Investigator — Bakırkoy Dr. Sadi Konuk Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arcoverde FVL, Andres MP, Borrelli GM, Barbosa PA, Abrao MS, Kho RM. Surgery for Endometriosis Improves Major Domains of Quality of Life: A Systematic Review and Meta-Analysis. J Minim Invasive Gynecol. 2019 Feb;26(2):266-278. doi: 10.1016/j.jmig.2018.09.774. Epub 2018 Sep 20. PMID 30244153